CLINICAL TRIAL: NCT07155369
Title: A Clinical Study Evaluating the Safety and Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA in Patients With Relapse/Refractory Autoimmune Diseases
Brief Title: UCAR T-cell Therapy Targeting CD19/ BCMA in Patients With Relapse/ Refractory Autoimmune Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Shanghai Xiniao Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-XZ-02
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus; Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCAR T-cell group (Experimental): Participants will receive the following interventions and dose escalated per protocol:
  Biological: UCAR-T cells Drug: Cyclophosphamide Drug: Fludarabine
  Interventions: Biological: UCAR-T cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: UCAR-T cells — UCAR-T cells will be administered intravenously as per the schedule specified in the protocol.
Drug: Cyclophosphamide — Cyclophosphamide will be administered intravenously.
Drug: Fludarabine — Fludarabine will be administered intravenously.

SUMMARY:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal allogeneic anti-CD19/BCMA CAR T-cells in With Relapse/Refractory Autoimmune Diseases.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy ofuniversal allogeneic anti-CD19/BCMA CAR T-cells in Patients With Relapse/Refractory Autoimmune Diseases.

Study intervention consists of a single infusion of universal allogeneic CART-cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old (inclusive), regardless of gender.
2. Positive expression of CD19 on peripheral blood B cells confirmed by flow cytometry.
3. Adequate hepatic, renal and bone marrow function.
4. Participants with relapsed or refractory autoimmune diseases, Including SLE or SSc.

Exclusion Criteria:

1. Participants with a history of severe drug allergies or allergic constitutions.
2. Presence or suspicion of uncontrolled or treatment-required fungal, bacterial, viral, or other infections.
3. Participants with insufficient cardiac function.
4. Participants with congenital immunoglobulin deficiencies.
5. History of malignancy within five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of UCAR T-cell in participants with relapse/ refractory autoimmune diseases | 2 years
  The incidence and severity of adverse events (AEs)
To evaluate the clinical responses and duration of UCAR-T cells in participants with relapse/ refractory autoimmune diseases | 2 years
  Proportion of participants achieving SRI-4 response, change in the Systemic Lupus Erythematosus Disease Activity Index(SLEDAI) from baseline

SECONDARY OUTCOMES:
To characterize the cellular kinetics of UCAR T-cell in participants with relapse/ refractory autoimmune diseases | 2 years
  AUC0-28d
To characterize the cellular kinetics of UCAR T-cell in participants with relapse/ refractory autoimmune diseases | 2 years
  Cmax
To characterize the cellular kinetics of UCAR T-cell in participants with relapse/ refractory autoimmune diseases | 2 years
  Tmax
To characterize pharmacodynamics of of UCAR-T cells in participants. | 2 years
  Changes in B-cell levels in the peripheral blood from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, China

IPD SHARING:
Plan to Share IPD: No